CLINICAL TRIAL: NCT00042185
Title: Austin Body Acceptance Study
Brief Title: Eating Disorder Prevention Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH061957 (NIH); R01MH061957 (NIH); DSIR 84-CTP
Record Dates: First submitted 2002-07-24; First posted 2002-07-26 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Eating Disorders
Keywords: Adolescence; Prevention and Control; Bulimia
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia

ARMS (4):
- Dissonance intervention (Experimental)
  Interventions: Behavioral: Dissonance Eating Disorder Prevention Program
- Healthy Weight Intervention (Active Comparator)
  Interventions: Behavioral: Healthy Weight Intervention
- Expressive writing control intervention (Active Comparator)
  Interventions: Behavioral: Expressive Writing Control Condition
- Assessment-only control condition (No Intervention)

INTERVENTIONS:
Behavioral: Dissonance Eating Disorder Prevention Program — In this intervention, participants voluntarily engaged in verbal, written, and behavioral exercises in which they critiqued the thin-ideal ideal. These exercises were conducted in sessions and in homework activities. For example, they wrote a counter-attitudinal essay about the costs associated with pursuit of the thin-ideal and engaged in a counter-attitudinal role-play in which they attempted to dissuade facilitators from pursuing the thin-ideal.
  Arms: Dissonance intervention
Behavioral: Healthy Weight Intervention — In this intervention, participants were encouraged to make gradual healthy and lasting changes to their diet and physical activity to balance their energy needs with their energy intake, and thereby achieve a healthier weight and body satisfaction. With support from the facilitator and group members, they initiated an individual lifestyle change plan to reduce intake of fat and sugar and to increase exercise using behavioral modification principles. Food and exercise diaries were used to identify behaviors to target in this lifestyle modification and to monitor change. Motivational enhancement activities were used to promote motivation for behavior change.
  Arms: Healthy Weight Intervention
Behavioral: Expressive Writing Control Condition — In this condition, which is based on the work of Pennebaker (1997), participants wrote about emotionally significant topics in three individual weekly 45-minute sessions. They were told that research indicates that body dissatisfaction is linked to emotional issues and that expressive writing helps resolve these issues. Sample topics included relationships or goals. They were told that their work would not be read and were asked to write continuously for the duration of the session about an emotionally important topic.
  Arms: Expressive writing control intervention

SUMMARY:
This study evaluated 2 eating disorder prevention programs designed to increase body satisfaction among adolescent females with body image concerns.

DETAILED DESCRIPTION:
Adolescent girls with body dissatisfaction (N=481; SD=1.4) were randomized to a dissonance-based thin-ideal internalization reduction program, healthy weight control program, expressive-writing control condition, or assessment-only control condition. Dissonance participants showed significantly greater decreases in thin-ideal internalization, body dissatisfaction, negative affect, eating disorder symptoms, and psychosocial impairment, and lower risk for eating pathology onset through 2-3 year follow-up than assessment-only controls. Dissonance participants showed greater decreases in thin-ideal internalization, body dissatisfaction, and psychosocial impairment than expressive-writing controls. Healthy weight participants showed greater decreases in thin-ideal internalization, body dissatisfaction, negative affect, eating disorder symptoms, and psychosocial impairment, less increases in weight, and lower risk for eating pathology and obesity onset through 2-3 year follow-up than assessment-only controls. Healthy weight participants showed greater decreases in thin-ideal internalization and weight than expressive writing controls. Dissonance participants showed a 60% reduction in risk for eating pathology onset and healthy weight participants showed a 61% reduction in risk for eating pathology onset and a 55% reduction in risk for obesity onset relative to assessment-only controls through 3-year follow-up, implying that the effects are clinically important and enduring.

ELIGIBILITY:
Inclusion criteria:

* Self-reported body image concerns

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 450
Dates: Start 2001-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Diagnostic Interview | 1 year

SECONDARY OUTCOMES:
The Ideal-Body Stereotype Scale-Revised, Satisfaction and Dissatisfaction with Body Parts Scale, Positive Affect and Negative Affect Scale-Revised | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- [Background] Stice E, Shaw H. Eating disorder prevention programs: a meta-analytic review. Psychol Bull. 2004 Mar;130(2):206-27. doi: 10.1037/0033-2909.130.2.206. PMID 14979770
- [Background] Stice E, Fisher M, Martinez E. Eating disorder diagnostic scale: additional evidence of reliability and validity. Psychol Assess. 2004 Mar;16(1):60-71. doi: 10.1037/1040-3590.16.1.60. PMID 15023093